CLINICAL TRIAL: NCT06462352
Title: Multicenter Study Comparing the Artificial Intelligence-Based Navicam Endoscopic Capsule With the Conventional Pillcam Endoscopic Capsule in Small Bowel Pathology
Brief Title: Multicenter Study Comparing AI-Based Navicam vs. Conventional Pillcam in Small Bowel Pathology
Acronym: NAVIPILL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Spanish Society of Digestive Endoscopy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: NAVIPILL
Record Dates: First submitted 2024-05-30; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-05

CONDITIONS: Small Intestine Disease
Keywords: capsule endoscopy; artificial intelligence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Navicam endoscopic capsule (Experimental): Navicam endoscopic capsule device for the study of small bowel pathology.
  Interventions: Device: Navicam SB capsule
- Pillcam endoscopic capsule (Active Comparator): Pillcam SB3 endoscopic capsule device for the study of small bowel pathology.
  Interventions: Device: Pillcam SB3

INTERVENTIONS:
Device: Navicam SB capsule — Exploration of the small bowel by Navicam SB endoscopic capsule.
  Arms: Navicam endoscopic capsule
Device: Pillcam SB3 — Exploration of the small bowel by Pillcam SB3 endoscopic capsule.
  Arms: Pillcam endoscopic capsule

SUMMARY:
Since its introduction in 2001, small bowel capsule endoscopy has been pivotal in diagnosing small bowel pathology due to its minimally invasive nature and high diagnostic accuracy. However, the technology has limitations, including prolonged reading times and the need for specialized endoscopists. The Navicam endoscopic capsule, leveraging artificial intelligence (AI) with ProScan™ for automated reading, promises to address these limitations by reducing reading times and enhancing diagnostic efficiency.

This study aims to assess the diagnostic concordance and to compare the efficiency of the AI-based Navicam capsule with the conventional Pillcam SB3 in the exploration of the small bowel.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, observational study involving multiple hospitals across Spain. At each site, patients will ingest both the Pillcam SB3 and Navicam capsules in a randomized order. Reading times, transit times, and diagnostic yield will be compared between the two devices. A central reading committee of experienced gastroenterologists will conduct blinded evaluations of both explorations using predefined criteria.

The primary endpoint is the diagnostic concordance between Navicam's AI-driven ProScan™ system and the conventional reading of Pillcam SB3, measured by Cohen's kappa index.

The secondary endpoints include to assess the correlation in lesion detection, video download times, gastric and small bowel transit times, total reading times, and adverse events.

The sample size is 147 patients, accounting for an expected 10% dropout rate, based on previous studies showing a diagnostic concordance kappa index of 0.6.

This study aims to establish that the AI-based Navicam capsule is at least as effective as the conventional Pillcam SB3 in diagnosing small bowel lesions, with potentially reduced reading times, thus enhancing clinical efficiency in small bowel diagnostics.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients over 18 years of age with any clinical indication to undergo a small bowel exploration using capsule endoscopy at the participating hospital.

Exclusion Criteria:

* Patients with known small bowel strictures detected by computed tomography (CT) or magnetic resonance imaging (MRI).
* Patients with a history of esophagogastric and small bowel surgery (excluding ileocecal resection).
* Patients with a clinical contraindication for small bowel capsule endoscopy.
* Hospitalized patients.
* Patients with pacemaker or Implantable Cardioverter Defibrillator (ICD).
* Patients scheduled for a MRI within 15 days after capsule endoscopy ingestion.
* Pregnant or actively breastfeeding patients.
* Patients with swallowing disorders requiring endoscopic placement of the capsule.
* Simultaneous participation in another clinical trial using any investigational drug or device.
* Concurrent life-threatening pathology or condition.
* Inability to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Concordance correlation coefficient in small bowel exploration (per-patient analysis) | From the start of recording up to 12 hours afterward
  To assess the concordance (k agreement) between Navicam (with ProscanTM AI-system) and Pillcam endoscopic capsule device in detecting patients with at least one significant small bowel lesion.

SECONDARY OUTCOMES:
Correlation coefficient in lesion detection (per-lesion analysis) | From the start of recording up to 12 hours afterward
  To assess the correlation between Navicam (AI-tool Proscan) and Pillcam in detecting small bowel lesions.
Reading time in minutes | From the start of recording up to 12 hours afterward
  To compare reading times of the small bowel between Navicam (Proscan) and Pillcam SB3.
Transit times in minutes | From the start of recording up to 12 hours afterward
  To compare gastric, small bowel, and colonic transit times between Navicam and Pillcam SB3.
Adverse events related to Navicam and/or Pillcam SB3 | From the start of recording up to 24 hours afterward
  Describe any adverse events during small bowel exploration.

CONTACTS AND LOCATIONS:
Overall Officials: Begoña González Suárez, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (16):
- Spain (16):
  - Hospital General Universitario Dr Balmis, Alicante
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Institut de Recerca Sant Pau (IR-Sant Pau), Barcelona
  - Hospital Universitario de Galdakao, Bilbao
  - Hospital General Universitario Virgen la Arrixaca, El Palmar
  - Hospital General Universitario de Elche, Elche
  - Hospital Clínico San Carlos, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital de Terrassa, Terrassa
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario i Politècnic La Fé, Valencia

IPD SHARING:
Plan to Share IPD: No